CLINICAL TRIAL: NCT01941186
Title: A Family Centered Intervention to Promote Optimal Child Development at the Interface of the Health System and Community
Brief Title: A Family Centered Intervention to Promote Optimal Child Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 13-010441
Record Dates: First submitted 2013-09-09; First posted 2013-09-13 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Developmental Delays
Keywords: Children; Developmental Delays; Early Intervention (EI); Patient Decision Aid (PDA)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Decision Aid (Experimental): After positive screen for a developmental concern the intervention group will receive the Patient Decision Aid (PDA), as well as, a text message reminder to follow up with Early Intervention.
  Interventions: Other: Patient Decision Aid
- Routine Care (No Intervention): After screening positive for a potential development delay those in the control arm will receive routine care, in this case, a handout explaining Early Intervention services.

INTERVENTIONS:
Other: Patient Decision Aid — Short informational video on developmental delays and early intervention services aimed at helping parents make an informed decision about whether to pursue early intervention services.
  Arms: Patient Decision Aid

SUMMARY:
This is a randomized controlled trial aimed at assessing the effectiveness of a patient decision aid (PDA) and text message reminder in promoting early intervention referral completion when infants and toddlers are identified with a developmental concern in the pediatric medical home. Subjects will be randomized to one of two study arms- (1) intervention (2) control condition. Subjects in the intervention arm will watch a video PDA and will receive a text message reminder approximately 7 to 14 business days after enrollment if they agree to the early intervention referral.

ELIGIBILITY:
Inclusion Criteria:

* Parent-child dyads in which the child is age 0 to 36 months screening positive for developmental concern and receiving care at a practice within Children's Hospital of Philadelphia Pediatric Research Consortium (PeRC).
* Caregivers able to give permission (informed consent).

Exclusion Criteria:

* Primary language other than English
* Children already enrolled in early intervention

Ages: 2 Days to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Manuel Jimenez, MD, MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 urban pediatric practice sites within the Children's Hospital of Philadelphia Pediatric Research Consortium, a primary care-based network including 31 practices in 2 states, between December 2013 and September 2014.
Pre-assignment Details: 164 parent-child dyads were assessed for eligibility and 100 were excluded. Reasons for exclusion were primarily because potential subjects either not meeting eligibility criteria (i.e., already received early intervention) or they declined to participate. 64 parent-child dyads were consented and randomized.
Groups:
- Patient Decision Aid: After positive screen for a developmental concern the intervention group received the Patient Decision Aid (PDA), as well as, a text message reminder to follow up with Early Intervention.
  Patient Decision Aid: Short informational video on developmental delays and early intervention services aimed at helping parents make an informed decision about whether to pursue early intervention services.
- Routine Care: After screening positive for a potential development delay those in the control received routine care, in this case, a handout explaining Early Intervention services.
Period: Randomization/Allocation to Study Group
Arm/Group | Patient Decision Aid | Routine Care
Started | 31 | 33
Completed | 31 | 33
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Patient Decision Aid | Routine Care
Started | 31 | 33
Completed | 30 | 33
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: 64 parent-child dyads were enrolled, randomized and included in the final analysis. 1 parent-child dyad who completed the intervention could not be contacted for follow-up to determine early intervention (EI) disposition within 1 year of enrollment. Intervention phase data was complete and is in the final analysis.
Groups:
- Routine Care: After screening positive for a potential development delay those in the control arm received routine care, in this case, a handout explaining Early Intervention services.
- Total: Total of all reporting groups
Arm/Group | Patient Decision Aid | Routine Care | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Customized [Number; unit: participants] — Child's Age
  participants
    Child: Age 1-12 months | 3 | 4 | 7
    Child: Age 13-24 months | 20 | 22 | 42
    Child: Age 25-36 months | 8 | 7 | 15
Age, Customized [Number; unit: participants] — Parent's Age
  participants
    Parent: 20 years and Under | 2 | 3 | 5
    Parent: 21-30 Years | 15 | 18 | 33
    Parent: 31-40 Years | 10 | 6 | 16
    Parent: Over 40 Years | 2 | 2 | 4
    Parent: Unknown Age | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Child's Gender
  Participants
    Female | 13 | 12 | 25
    Male | 18 | 21 | 39
Sex: Female, Male [Count of Participants; unit: Participants] — Parent's Gender
  Participants
    Female | 5 | 5 | 10
    Male | 26 | 28 | 54
Race/Ethnicity, Customized [Number; unit: participants] — Parent's Race
  participants
    Black/African American | 24 | 32 | 56
    Other | 7 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64
Parent's Education [Number; unit: participants]
  Less than High School | 1 | 4 | 5
  High School Graduate | 23 | 27 | 50
  Post Secondary Education | 7 | 2 | 9
Parent's Employment Status [Number; unit: participants]
  Employed | 17 | 20 | 37
  Unemployed | 14 | 13 | 27
Parent's Marital Status [Number; unit: participants]
  Married/Living with Partner | 13 | 13 | 26
  Divorced/Separated | 4 | 2 | 6
  Never Married | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Number of Participants Who Completed Early Intervention Intake and Evaluation Visits Between Treatment Groups
Description: Completed intake and evaluation by the early intervention (EI) agency was assessed by parent report and by chart review. A member of the study team contacted parents within 6 months of the first study visit to obtain this information. Additionally, a chart review seeking written feedback information regarding referral disposition from the EI agency was completed.
Time Frame: Up to 1 year after randomization
Population: One parent-child dyad had missing information regarding EI intake and evaluation. Given the absence of information on referral outcome, this parent-child dyad was included in the final evaluation as having not received an EI intake and evaluation.
Measure: Number; unit: participants
Arm/Group | Patient Decision Aid | Routine Care
Number analyzed (Participants) | 31 | 33
participants
  Early Intervention Intake | 20 | 21
  Early Intervention Evaluation | 17 | 17

2. Secondary Outcome: Change in Parental Knowledge and Attitudes From Pre- to Post-Intervention
Description: Pre and post knowledge and attitudes regarding developmental delay and early intervention (EI) were assessed by asking participants to respond to 14 statements using a 6 point Likert scale that ranged from strongly disagree to strongly agree. Questions mapped to the video decision aid content viewed by participants. Participants in the intervention arm completed the questions before and after watching the video and participants in the control arm completed the questions sequentially. Secondary outcome measures assessed in the survey included Parent Uncertainty About Early Intervention and Parental Predisposition for Early Intervention.
Time Frame: Up to 7 days
Population: All parent-child dyads who were enrolled and randomized were included in the analysis.
Measure: Number; unit: percentage of participants
Groups:
- Patient Decision Aid: Strongly Disagree; Routine Care: Strongly Disagree: Percentage of parents who answered "strongly disagree" to questions during pre and post intervention
- Patient Decision Aid: Disagree; Routine Care: Disagree: Percentage of parents who answered "disagree" to questions during pre and post intervention
- Patient Decision Aid: Somewhat Disagree: Percentage of parents who answered "somewhat disagree" to questions during pre and post
- Patient Decision Aid: Somewhat Agree; Routine Care: Somewhat Agree: Percentage of parents who answered "somewhat agree" to questions during pre and post intervention
- Patient Decision Aid: Agree; Routine Care: Agree: Percentage of parents who answered "agree" to questions during pre and post intervention
- Patient Decision Aid: Strongly Agree; Routine Care: Strongly Agree: Percentage of parents who answered "Strongly Agree" to questions during pre and post intervention
- Routine Care: Somewhat Disagree: Percentage of parents who answered "somewhat disagree" to questions during pre and post intervention
Arm/Group | Patient Decision Aid: Strongly Disagree | Patient Decision Aid: Disagree | Patient Decision Aid: Somewhat Disagree | Patient Decision Aid: Somewhat Agree | Patient Decision Aid: Agree | Patient Decision Aid: Strongly Agree | Routine Care: Strongly Disagree | Routine Care: Disagree | Routine Care: Somewhat Disagree | Routine Care: Somewhat Agree | Routine Care: Agree | Routine Care: Strongly Agree
Number analyzed (Participants) | 31 | 31 | 31 | 31 | 31 | 31 | 33 | 33 | 33 | 33 | 33 | 33
percentage of participants
  All learn to talk, walk, think @ same time (pre) | 48 | 35 | 6 | 10 | 0 | 0 | 52 | 33 | 9 | 3 | 0 | 3
  All learn to talk, walk, think @ same time (post) | 42 | 35 | 3 | 6 | 3 | 9 | 52 | 30 | 9 | 6 | 3 | 0
  Longer to talk, walk, think may be delayed (pre) | 10 | 32 | 10 | 23 | 19 | 6 | 9 | 33 | 21 | 21 | 6 | 9
  Longer to talk, walk, think may be delayed (post) | 10 | 10 | 10 | 23 | 35 | 13 | 15 | 30 | 12 | 33 | 6 | 3
  All with delays get better on their own (pre) | 19 | 29 | 6 | 19 | 19 | 6 | 3 | 30 | 15 | 30 | 15 | 6
  All with delays get better on their own (post) | 16 | 39 | 10 | 29 | 3 | 3 | 18 | 21 | 21 | 24 | 9 | 6
  Behavior/Learning probs in school w/o help (pre) | 10 | 16 | 6 | 26 | 29 | 13 | 6 | 9 | 12 | 30 | 27 | 15
  Behavior/Learning probs in school w/o help (post) | 3 | 3 | 6 | 13 | 45 | 29 | 3 | 0 | 15 | 30 | 30 | 21
  Know more about child's develop than others (pre) | 10 | 10 | 10 | 19 | 19 | 32 | 6 | 24 | 12 | 33 | 15 | 9
  Know more about child's develop than others (post) | 10 | 6 | 6 | 29 | 29 | 19 | 6 | 12 | 15 | 24 | 27 | 15
  If delayed want to work with child on my own (pre) | 23 | 39 | 10 | 10 | 16 | 3 | 9 | 27 | 24 | 18 | 21 | 0
  If delayed want to work with child on my own (pos) | 23 | 35 | 16 | 16 | 3 | 6 | 6 | 27 | 21 | 9 | 18 | 18
  EI helps kids w/develop delay (pre) | 6 | 0 | 0 | 16 | 42 | 35 | 0 | 0 | 0 | 9 | 64 | 27
  EI helps kids w/develop delay (post) | 3 | 0 | 0 | 13 | 42 | 42 | 0 | 0 | 0 | 18 | 48 | 33
  You have to pay for EI services (pre) | 23 | 45 | 13 | 13 | 6 | 0 | 27 | 39 | 21 | 6 | 6 | 0
  You have to pay for EI services (post) | 55 | 35 | 0 | 6 | 3 | 0 | 39 | 45 | 9 | 3 | 3 | 0
  EI services can be in home or daycare (pre) | 6 | 3 | 3 | 6 | 51 | 29 | 0 | 0 | 3 | 6 | 48 | 42
  EI services can be in home or daycare (post) | 3 | 3 | 0 | 6 | 35 | 52 | 0 | 0 | 0 | 15 | 45 | 39
  EI provider must come to home (pre) | 13 | 16 | 16 | 23 | 19 | 13 | 9 | 36 | 18 | 15 | 12 | 9
  EI provider must come to home (post) | 10 | 23 | 10 | 23 | 23 | 13 | 12 | 7 | 15 | 21 | 18 | 6
  Once EI starts you cannot stop (pre) | 32 | 35 | 16 | 3 | 13 | 0 | 45 | 36 | 6 | 3 | 3 | 6
  Once EI starts you cannot stop (post) | 48 | 32 | 6 | 6 | 3 | 3 | 39 | 42 | 9 | 0 | 6 | 3
  Studies show EI helps make progress (pre) | 6 | 3 | 0 | 13 | 45 | 32 | 0 | 0 | 6 | 18 | 58 | 18
  Studies show EI helps make progress (post) | 3 | 0 | 0 | 10 | 42 | 45 | 0 | 0 | 6 | 9 | 58 | 27
  Resources like EI can help my family & I (pre) | 6 | 0 | 3 | 13 | 35 | 42 | 0 | 0 | 0 | 9 | 52 | 39
  Resources like EI can help my family & I (post) | 3 | 0 | 0 | 10 | 35 | 52 | 0 | 0 | 0 | 12 | 58 | 30
  I'm comfortable with EI staff in my home (pre) | 6 | 3 | 3 | 16 | 29 | 42 | 0 | 3 | 3 | 12 | 48 | 33
  I'm comfortable w/EI staff in my home (post) | 3 | 0 | 6 | 10 | 39 | 42 | 0 | 0 | 6 | 12 | 45 | 36

3. Other Pre Specified Outcome: Parent Uncertainty About Early Intervention
Description: Parental uncertainty about whether to enroll their child in Early Intervention will be evaluated using a survey.
Time Frame: Up to 7 days
Population: All survey data is presented collectively in Secondary Outcome Measure, "Change in Parental Knowledge and Attitudes From Pre- to Post-Intervention". A separate analysis was not completed.
Arm/Group | Patient Decision Aid | Routine Care
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Parental Predisposition for Early Intervention
Description: Parental predisposition for early intervention services will be measured using surveys.
Time Frame: Up to 7 days
Population: as for outcome 3
Arm/Group | Patient Decision Aid | Routine Care
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Feasibility of the Patient Decision Aid
Description: The feasibility of the patient decision aid (PDA) will be measured by calculating the number of individuals who refuse to participate, time that it takes to complete the PDA, and the number of patients who complete the Early Intervention referral.
Time Frame: Up to 7 days
Population: Data was not collected regarding the time to complete PDA and/or number of Early Intervention referrals for the total population, thus data for this outcome measure was not able to be analyzed as outlined at the time of protocol development.
Arm/Group | Patient Decision Aid | Routine Care
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Acceptability of the Patient Decision Aid for Early Intervention Referral
Description: The acceptability of using the patient decision aid for early intervention will be assessed by having patients and providers complete surveys on the intervention.
Time Frame: Up to 7 days
Population: Provider information was not collected as outlined in the initial protocol design. All survey data is presented collectively in Secondary Outcome Measure, "Change in Parental Knowledge and Attitudes From Pre- to Post-Intervention". This includes elements of parent acceptability. A separate analysis was not completed.
Arm/Group | Patient Decision Aid | Routine Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the duration of participation (up to 1 year)
Arm/Group | Patient Decision Aid | Routine Care
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

LIMITATIONS AND CAVEATS:
Given that the study recruited a convenience sample from one primary care network, findings may not be generalizable to all settings. Also worth noting, EI services differ by state and some of the information is not applicable in all states.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes